CLINICAL TRIAL: NCT07123766
Title: A Prospective, Multicenter, Single-Arm Study With Objective Performance Criteria Evaluating the Efficacy and Safety of PoliaValve® Artificial Heart Valve
Brief Title: Clinical Investigation for the PoliaValve Aortic Heart Valve- India
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Hearthill Medical Technology Co.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PoliaValve-SA-03
Record Dates: First submitted 2025-07-28; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: AORTIC VALVE DISEASES; Aortic Valve Stenosis; Aortic Valve Regurgitation
Keywords: Heart Valve Diseases; Aortic Valve Regurgitation; Aortic Valve Disease; Polymeric Aortic Valve
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group(PoliaValve) (Experimental): Patients receiving the PoliaValve (Aortic) from HearrHill Medical
  Interventions: Device: PoliaValve (Aortic)

INTERVENTIONS:
Device: PoliaValve (Aortic) — Aortic Valve Replacement

SUMMARY:
The purpose of this study is to conduct a clinical investigation of the HeartHill PoliaValve Aortic Valve to collect evidence on the device's safety and performance.

DETAILED DESCRIPTION:
The PoliaValve is indicated as a replacement for diseased, damaged, or malfunctioning native aortic heart valve via open heart surgery. The study is a single-arm, open label, non-randomized multi- center clinical trial. Up to 10 sites in the country of India will enroll up to 50 patients. These patients will follow the study schedule for 1 year after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Is 45 years or older
* Provide written informed consent prior to trial procedures after standard of care studies and tests indicate that the patient needs aortic valve replacement
* Agrees to attend all follow-up assessments for up to 1 year and is willing to comply with specified follow-up evaluations for the clinical trial
* Diagnosed with severe symptomatic aortic valve stenosis and/or regurgitation

Exclusion Criteria:

* Requires multiple valve replacement / repair
* Requires emergency surgery
* Has had prior valve surgery
* Requires a surgical procedure outside of the cardiac area
* Requires a cardiac procedure other than a CABG or root enlargement or aortic root replacement
* Requires or are planning another unrelated surgery within 12 months of undergoing implantation of the study device
* Has active endocarditis/myocarditis or within 3 months to the scheduled surgery
* Has renal insufficiency as determined by creatinine (S-Cr) level as ≥ 1.5 mg/dl or end-stage renal disease requiring chronic dialysis at screening visit
* Has MRI or CT scan confirmed stroke, cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 3 months (90 days) prior to planned valve surgery
* Has acute myocardial infarction (AMI) within 30 days prior to planned valve surgery
* Has life expectancy to less than 12 months
* Diagnosed with hypertrophic obstructive cardiomyopathy (HOCM), except patients who have isolated subaortic muscular hypertrophy diagnosed at the time of surgery
* Diagnosed with abnormal calcium metabolism and/or hyperparathyroidism
* Echocardiographic left ventricular ejection fraction <25%
* Echocardiographic evidence of an intra-cardiac thrombus or vegetation
* Hemodynamic or respiratory instability requiring inotropic support, mechanical circulatory support, or mechanical ventilation within 30 days prior to planned valve surgery
* Documented leukopenia (WBC < 4.0 x 103/µL), acute anemia (Hgb < 10.0 gm/dl or 6 mmol/L), thrombocytopenia (platelet count < 100 x103/µL) or history of bleeding diathesis or coagulopathy
* Has prior organ transplant or is currently an organ transplant candidate
* Current or recent participation (within 6 weeks prior to surgery) in another drug or device trial
* Pregnant, lactating or planning to become pregnant during the duration of participation in trial
* Currently incarcerated or unable to give voluntary informed consent
* Documented history of substance (drug or alcohol) abuse within the last 5 years prior to implant
* Requires concomitant left ventricular assist device (LVAD) placement, Impella placement, and/or intra-aortic balloon pump
* Currently has uncontrolled infection
* Currently diagnosed as uncontrolled diabetes mellitus (Random BLS > 300 mg/dl)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Clinical Outcomes Events | 12 months following patient enrollment completion
  The rate of adverse events will be compared to clinical outcomes for surgically implanted heart valves reported in the literature: a) thromboembolism, b) valve thrombosis, c) major paravalvular leak, d) major hemorrhage, e) endocarditis, f) all-caused death, g) valve related death, h) valve related reoperation, i) valve explant, j) hemorrhage, k) all-cause reoperation

SECONDARY OUTCOMES:
Effective Orifice Area (EOA) | 12 months following patient enrollment completion
  Using doppler echocardiography to Measure Effective Orifice Area (EOA)
Mean Pressure Gradient(MPG) | 12 months following patient enrollment completion
  The mean pressure gradient (MPG) is a measure of the average pressure difference across a valve or a specific area in a fluid system, often measured by transthoracic echocardiogram.
New York Heart Association(NYHA) Improvement Assessment | 12 months following patient enrollment completion
  Clinically significant improvement (one grade) in the New York Heart Association (NYHA) functional classification status at 365 days compared to baseline. a. Class I - No symptoms and no limitations in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc. b. Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity. c. Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100m). Comfortable only at rest. d. Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Rate of Stroke | 12 months following patient enrollment completion
  Assessment of patient experiencing a stroke verified by imaging and or physical exam
Rate of Transient Ischemic Attack(TIA) | 12 months following patient enrollment completion
  Assessment of patient having a transient ischemic attack(TIA) verified by imaging and or physical exam
Intensive Care Unit(ICU) Duration of Stay | 30 days post procedure
  Length of stay in the ICU post valve implantation defined as arrival time/date in hours and minutes to transfer to floor time/date in hours and minutes.
Ventilation Time | 30 days post procedure
  Ventilation time in hours defined as arrival time/date in recovery in hours and minutes to date and time extubated in hours and minutes
Rate of New Onset Atrial Fibrillation | 12 months post procedure
Length of Stay in Hospital | 30 days post procedure
Readmission | 30 days post procedure
  Patient readmission to the hospital post discharge measured by date/time
Hemolysis screen | 12 months post procedure
  Hemolysis screen is measured by blood tests including hemoglobin and liver enzyme assessments

IPD SHARING:
Plan to Share IPD: No